CLINICAL TRIAL: NCT03673436
Title: Effect of Lumbar Spinal Fusion Predicted by Physiotherapists: A Prospective Cohort Study
Brief Title: Effect of Lumbar Spinal Fusion Predicted by Physiotherapists
Status: Completed | Type: Observational
Sponsor: Rigshospitalet, Denmark (Other)
Collaborators: Frederiksberg University Hospital (Other)
Responsible Party: Principal Investigator, Heidi Tegner, Clinical physiotherapy supervisor, PT, MScH, Rigshospitalet, Denmark
Other Study IDs: 1
Record Dates: First submitted 2018-09-12; First posted 2018-09-17 (Actual); Last update posted 2021-03-10 (Actual); Status verified 2021-03

CONDITIONS: Low Back Pain
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with low back pain: Cohort of 200 low back pain patients, 18 years+, who have been undergoing a lumbar spinal fusion
  Interventions: Procedure: Lumbar spinal fusion

INTERVENTIONS:
Procedure: Lumbar spinal fusion — The patient got a instrumented fusion of a maximum of 3 adjacent vertebrae

SUMMARY:
The main purpose of this study is to investigate if improvements in patient self-reported pain, symptoms, function and quality of life 12 months after Lumbar spinal fusion among patients that have good projected prognosis differ from those among patients with a poor projected prognosis.

The secondary purpose is to explore the underlying factors of the physiotherapists projected prognosis to identify objective and possible modifiable candidate prognostic factors for recovery.

DETAILED DESCRIPTION:
Background:

Over recent decades, an increasing number of patients with Chronic Low Back Pain (CLBP) undergo surgical lumbar spinal fusion (LSF). For many of the patients LSF is their last resort in the hope of a better life with less pain, disability and use of medication. Unfortunately, several reports show, that the pain level remains the same after LSF for many patients, and that consumption of medication remains unchanged in almost 50 % of the patients.

Knowing that characteristics such as maladaptive coping strategies, fear avoidance beliefs and pain catastrophizing seem to be predictive of worse outcome in pain, function and quality of life after surgery. It is important to assess how these individual factors in the postsurgical rehabilitation can be addressed.

The single physiotherapists have an essential role in mobilizing the LSF patient post-operatively. In clinical practice it is not enough for the physiotherapists to use their biomechanical understanding of LSF material and heeling processes, it is also essential to use a so-called "silent knowledge" of experience and personal interaction with the patient.

It remains unknown if this "silent knowledge" is a reliable predictor of the outcome of LSF surgery. If the physiotherapist can predict the outcome, it is important to explore which factors the physiotherapist rely their prognosis upon in order to identify objective and possible modifiable candidate prognostic factors for recovery.

The aim of this study is to assess if physiotherapists attending inpatients at public back surgery hospitals can predict the future course (post hospitalisation) of recovery of patients undergoing LSF. The study will also break down the physiotherapists' "silent knowledge" in an attempt to identify objective (and hopefully modifiable) candidate prognostic markers of recovery.

ELIGIBILITY:
Inclusion Criteria:

* Received primary LSF surgery for treatment of CLBP
* Degenerative lumbar disease with or without lumbar spondylolisthesis grades 1 to 2
* Fusion of a maximum of 3 adjacent vertebrae
* Above 18 years of age
* Competence in the Danish language
* Has an email address

Exclusion Criteria:

* Prior LSF surgery
* Cognitive impairments that preclude reliable answers to patient reported outcome questionnaire

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population consist of 200 patients with lumbar spinal fusion operated at a hospital in Denmark
Sampling Method: Probability Sample
Enrollment: 202 (Actual)
Dates: Start 2018-09-30 (Actual); Primary Completion 2020-10-01 (Actual); Study Completion 2020-10-01 (Actual)

PRIMARY OUTCOMES:
Oswestry Disability Index | 1 year
  Disability will be measured using the Oswestry Disability Index. ODI is a validated measure of condition-specific disability originally developed for patients with LBP. The ODI consists of ten items regarding pain intensity, personal care, lifting, walking, sitting, standing, sleeping, sex life, social life, and traveling. For each item the patient chooses one of six answers, with 0 representing no difficulty in the activity and 5 representing maximal difficulty.

SECONDARY OUTCOMES:
Patient reported movement capacity | 1 year
  Patients are asked to mark the position along a horizontal 10-cm line that best corresponded to their movement capacity. The endings of the line have verbal descriptions: 0 (''very poor capacity'') - 100 ("very good capacity")
Back Pain | 1 year
  A visual analogue scale (VAS) is a simple and frequently used method for the assessment of variations in intensity of pain. Patients are asked to mark the position along a horizontal 10-cm line that best corresponded to their pain intensity. The endings of the line have verbal descriptions: 0 (''no pain'') - 100 ("the worst pain imaginable")
Leg Pain | 1 year
  A visual analogue scale (VAS) is a simple and frequently used method for the assessment of variations in intensity of pain. Patients are asked to mark the position along a horizontal 10-cm line that best corresponded to their pain intensity. The endings of the line have verbal descriptions: 0 (''no pain'') - 100 ("the worst pain imaginable")
Health outcome and quality of life | 1 year
  Quality of life will be assessed using the EuroQol 5 Dimensions 3 levels (EQ-5D-3L). The EQ-5D is a generic questionnaire developed by an international research group including re-searchers from Denmark. EQ-5D-3L consist of 5 dimensions in health-related quality of life: Mobility, Self-care, usual activities, Pain/discomfort, and anxiety/depression. Each dimension is divided into three levels: no problems, some problems or extreme problems. EQ-5D-3L also include a 20-cm vertical scale, were the respondent are asked to describe his/her own health with endpoints of 'best imaginable health state' set at 100 and 'worst imaginable health state' set at 0. The EQ-5D has been validated in Danish, including the development of preference values and Danish population norms.
Questionnaire regarding postoperative rehabilitation | 1 year
  We will administer a questionnaire that includes questions regarding the postoperative rehabilitation. It is questions regarding: setting, duration, participation and the degree of relevance to the individual patient. The patient will answer the questionnaire by a yes or no and detailed answers by text.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Occupational and Physiotherapy, Rigshospitalet Glostrup, Glostrup Municipality, Denmark

IPD SHARING:
Plan to Share IPD: Undecided